CLINICAL TRIAL: NCT05918588
Title: A Phase 1, Placebo-Controlled, Double-Blind, Dose-Escalating Study to Examine the Safety and Tolerability of Multiple Doses of KD025 (Formerly Called SLX-2119) in Healthy Male and Post- Menopausal Female Subjects
Brief Title: A Study to Determine the Effect of Multiple Oral Doses and Regimens of KD025 in Healthy Male and Post-menopausal Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kadmon, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: KD025-102; U1111-1290-9646 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Immune System Disorder (Healthy Volunteer)
MeSH Terms: conditions — Immune System Diseases | interventions — KD025

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental): 500 mg KD025 or placebo once daily (QD) for 7 days
  Interventions: Drug: Belumosudil mesylate; Drug: Placebo
- Cohort 2 (Experimental): 800 mg KD025 or placebo QD for 7 days
  Interventions: Drug: Belumosudil mesylate; Drug: Placebo
- Cohort 3 (Experimental): 500 mg KD025 or placebo twice daily (BID) for 7 days
  Interventions: Drug: Belumosudil mesylate; Drug: Placebo
- Cohort 4 (Experimental): 1000 mg KD025 or placebo QD for 7 days
  Interventions: Drug: Belumosudil mesylate; Drug: Placebo

INTERVENTIONS:
Drug: Belumosudil mesylate — Pharmaceutical form: capsule; Route of administration: oral
  Other Names: KD025; SAR445761
Drug: Placebo — Pharmaceutical form: capsule; Route of administration: oral

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and pharmacokinetics of multiple oral doses and regimens of KD025 in healthy male and post-menopausal female participants.

DETAILED DESCRIPTION:
Up to approximately 37 days including safety follow up period of 30 days after participant is treated with the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants between the ages of 18 and 55 years, inclusive.
* Female who was not of reproductive potential.
* Able to provide written informed consent prior to the performance of any study specific procedures.
* Body mass index (BMI) range of 19-30 kilogram per square meter (kg/m2), inclusive.

Exclusion Criteria:

* Past or present disease that is judged by the investigator to have the potential to interfere with the study procedures, compromise safety, or affect the PK evaluations.
* Known sensitivity to Rho-associated coiled-coil containing serine/threonine protein kinases (ROCK2) inhibitor agents or to any of the constituents of the KD025 formulation.

The above information is not intended to contain all considerations relevant to the potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2013-11-21 (Actual); Primary Completion 2014-03-06 (Actual); Study Completion 2014-03-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events and serious adverse events | Up to approximately 37 days
  Safety observations and measurements include AEs, safety laboratory tests, vital sign measurements, physical examinations, and ECGs.

SECONDARY OUTCOMES:
Cmax of KD025 and its metabolites [M1 (KD025m1) and M2 (KD025m2)] | Predose and multiple timepoints up to 48 hours postdose on Days 1 and 7
  Cmax is maximum plasma concentration determined directly from the concentration time profile
tmax of KD025 and its metabolites [M1 (KD025m1) and M2 (KD025m2)] | Predose and multiple timepoints up to 48 hours postdose on Days 1 and 7
  tmax is observed time to reach peak plasma concentration
AUC0-24 of KD025 and its metabolites [M1 (KD025m1) and M2 (KD025m2)] | Predose and multiple timepoints up to 48 hours postdose on Days 1 and 7
  AUC0-24 is area under the plasma concentration-time curve from predose (time 0) to 24 hours Postdose
AUCinf of KD025 and its metabolites [M1 (KD025m1) and M2 (KD025m2)] | Predose and multiple timepoints up to 48 hours postdose on Days 1 and 7
  AUCinf is area under the concentration-time curve from predose (time 0) extrapolated to Infinity
Cmin of KD025 and its metabolites [M1 (KD025m1) and M2 (KD025m2)] | Predose and multiple timepoints up to 48 hours postdose on Days 1 and 7
  Cmin is minimum or "trough" plasma concentration after its administration and just prior to the administration of a subsequent dose as determined from the concentration time profile
t1/2 of KD025 and its metabolites [M1 (KD025m1) and M2 (KD025m2)] | Predose and multiple timepoints up to 48 hours postdose on Days 1 and 7
  t1/2 is terminal elimination half-life

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational site, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org